CLINICAL TRIAL: NCT04007978
Title: Efficacy and Safety of Anti-CD22 CAR-T Therapy in Patients With Relapsed/Refractory B-cell Malignancies: a Single-center, Open-label, Single-arm Clinical Study
Brief Title: Anti-CD22 Chimeric Antigen Receptor (CAR)-Modified T Cell Therapy for Relapsed Refractory B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Bio-Raid Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-CART-CD22-01
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: B Cell Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Third generation CAR-T cells (Experimental): Patients receive CD22 CAR-T cells transduced with a lentiviral vector on day 0 in the absence of disease progression or unacceptable toxicity.
  Interventions: Genetic: Third generation CAR-T cells

INTERVENTIONS:
Genetic: Third generation CAR-T cells — Patients receive CD22 CAR-T cells transduced with a lentiviral vector on day 0 in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of anti-CD22 CAR-T cells in patients with relapsed or refractory B-cell Malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells (CAR-T cells) have the capabilities to recognize tumor associated antigen and kill tumor cells specifically. CAR-T therapy showed great effect on patients with relapsed or refractory B-cell malignancies. CAR consists of single chain variable fragment (scFv) and activation domain of T cell. In preclinical study, the researchers constructed a third generation CAR containing CD137 and CD28 costimulatory domains.

This study aims to evaluate the safety and effectiveness of anti-CD22 CAR-T cells in patients with relapsed or refractory B-cell Malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.
2. Male or female patients aged 14 to 70 years (including 14 and 70 years old).
3. Pathological and histological examination confirmed CD22+ B-cell malignancies, and patients met the following criteria for refractory or relapsed B-cell malignancies.

   A.Refractory/relapsed B-cell lymphoblastic leukemia (Meeting one of the following)

   i. Recurrence within 6 months after first remission.

   ii. Primary refractory disease which cannnot achieve complete remission (CR) after 2 cycles of standardized chemotherapy regimen.

   iii. Failure to achieve CR or relapse after one line or multiple lines of salvage chemotherapy.

   iv. Not suitable for hematopoietic stem cell transplantation (HSCT), or abandon HSCT due to various restrictions, or relapse after HSCT.

   B.Refractory/relapsed B-cell lymphoma (Meeting 1 of the first 4 items plus item 5)

   i. Tumor shrinkage less than 50% or disease progression after 4 cycles of standard chemotherapy.

   ii. Achieved CR after standard chemotherapy, but relapsed within 6 months.

   iii. 2 or more relapses after CR.

   iv. Not suitable for HSCT, or abandon HSCT due to various restrictions, or relapse after HSCT.

   v. Subjects must have received adequate treatment in the past, including anti-CD20 monoclonal antibody and combination chemotherapy with anthracyclines.
4. B-cell malignancies include the following three types

   A. B-cell acute lymphoblastic leukemia (B-ALL)

   B. Indolent B-cell lymphoma (CLL, FL, MZL, LPL, HCL)

   C. Invasive B-cell lymphoma (DLBCL, BL, MCL)
5. Having a measurable or evaluable lesion

   A. Patients with lymphoma require a single lesion≥15mm or 2 or more lesions≥10mm.

   B. Patients with leukemia require persistent positive or positive relapse of bone marrow MRD.
6. Patient's main organs functioning well

   A. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin≤34.2μmol/L

   B. Renal function: Creatinine < 220μmol/L.

   C. Pulmonary function: Indoor oxygen saturation≥95%.

   D. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥40%.
7. The patients did not receive any antitumor treatments such as chemotherapy, radiotherapy and immunotherapy (such as immunosuppressive drugs) within 4 weeks before enrollment, and the toxicity related to previous treatments had returned to < 1 level at enrollment (except for low grade toxicity such as alopecia).
8. The patient's peripheral superficial venous blood flow smoothly, which can meet the needs of intravenous drip.
9. Patient ECOG score≤ 2, estimated survival time≥3 months.

Exclusion Criteria:

1. Have a history of epilepsy or other central nervous system diseases.
2. Women who are pregnant (urine/blood pregnancy test positive) or lactating.
3. Male or female with a pregnancy plan in the next 1 year.
4. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 year after enrollment.
5. Uncontrolled infectious disease within 4 weeks prior to enrollment.
6. Active hepatitis B/C virus infection.
7. HIV infected patients.
8. Suffering from a serious autoimmune disease or immunodeficiency disease.
9. The patient is allergic to macromolecular biopharmaceuticals such as antibodies or cytokines.
10. The patient participated in other clinical trials within 6 weeks prior to enrollment.
11. Systemic use of corticosteroids within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids).
12. Suffering from mental diseases.
13. Patient has drug abuse/addiction.
14. According to the researcher's judgment, the patient has other unsuitable enrollment conditions.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 3 years
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
One-month remission rate | 1 month
  Response of B-ALL to CAR-T therapy was assessed on day 30 (±2), against the National Comprehensive Cancer Network (NCCN, Version 1.2015).
Overall survival | 3 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up (censored).
Event-free survival | 3 years
  EFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 3 years
  RFS was calculated from the first CAR-T cell infusion to relapse or last visit (censored).
Rate of anti-CD22 CAR-T cells in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) rate of CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD22 CAR-T cells in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD22 CAR copies in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of anti-CD22 CAR copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No